CLINICAL TRIAL: NCT02637102
Title: The UK CArdiac and Vascular Surgery Interventional Anaemia Response Study: An Observational Cohort Study to Determine the Impact and Effect of Anaemia in Patients Awaiting Vascular and Cardiac Surgery
Brief Title: The UK CAVIAR Study
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0659
Record Dates: First submitted 2015-11-27; First posted 2015-12-22 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Iron Deficiency; Cardiac Patients; Anaemia; Vascular Patients
MeSH Terms: conditions — Iron Deficiencies; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing cardiac or vascular surgery
  Interventions: Other: Not applicable - observational study

INTERVENTIONS:
Other: Not applicable - observational study

SUMMARY:
CAVIAR is a multicentre prospective observational study. Centres for cardiac and vascular surgery assess and manage patients in different ways before surgery. Some centres have introduced the use of intravenous iron therapy for patients with anaemia in the preoperative setting. Consequently regional variation exists in the assessment and management of patients before cardiac and vascular surgery. We aim to observe and measure these differing pathways and observe if there is variation in iron deficiency and anaemia and the impact of these variables on patient cardiorespiratory function as well as post-operative outcomes.

[Sub-Study] For patients who are receiving intravenous iron therapy as part of their routine clinical care, we wish to observe this effect in more detail. We will assess the impact of the treatment on well-being, blood count and fitness. Information will be collected through Quality of Life questionnaires, total haemoglobin mass test (via blood collection) and fitness testing.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 18 years or older
2. Screening [Hb] < 120 g/L (for females) or < 130g/L (for males)
3. Undergoing elective cardiac OR vascular surgery:

   * Coronary artery bypass (CABG), or valvular surgery, or combined CABG and valve surgery.
   * Repair or replacement of thoracic or abdominal aorta (open or endovascular).
4. Able to provide informed consent
5. (if applicable) Able to perform CPET or 6MWT if consented to take part in the sub study

Exclusion Criteria:

1. Pregnancy or lactation
2. Adults with known underlying history of learning disabilities, or adults who do not have mental capacity to consent for themselves
3. Prisoners
4. Renal dialysis (current or planned within the next 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring major cardiac or vascular surgery will be identified from routine clinical care. Most patients are routinely referred for pre-operative assessment, although local protocols vary between centres. Assesments at the pre-operative assessment clinic (PAC) may include (but not limited to) routine blood tests (full blood count, urea and electrolytes, etc.), history and examination, cardiorespiratory fitness assessment by 6 minute walk test (6MWT) or cardiopulmonary exercise testing (CPET). In some centres, patients with anaemia will receive intravenous iron at PAC or in a separate anaemia clinic.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2015-11; Primary Completion 2018-03 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in Haemoglobin | From baseline to before surgery (within 10-42 days)

SECONDARY OUTCOMES:
Changes in biomarkers of iron deficiency (e.g. hepcidin, ferritin, TfSats) | From baseline to after IV iron (within 4-6 weeks before surgery)
Haemoglobin | Before surgery (within 10-42 days) to post surgery (within 3 weeks)
Unit of blood transfused | Hospital stay (within 7 days)
ICU and hospital length of stay | Within 30 days
Renal function (change in creatinine) | From baseline to before surgery (within 10-42 days)
Renal function (change in creatinine) | From baseline to post surgery (within 3 weeks)
Complications | Within 30 days post surgery
Feasibility - number of successful patient recruitment and consent | Within a year
Total haemoglobin mass test (Sub-study ONLY) | From baseline to after IV iron (within 4-6 weeks before surgery)
Functional exercise testing (CPET or 6MWT) (Sub-study ONLY) | From baseline to after IV iron (within 4-6 weeks before surgery)
Quality of Life (Sub-Study ONLY) | From baseline to i) after IV iron (within 4-6 weeks before surgery), ii) post surgery (within 3 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Toby Richards, MD FRCS, Principal Investigator — University College, London

REFERENCES:
- [Derived] Chau M, Richards T, Evans C, Butcher A, Collier T, Klein A. The UK Cardiac and Vascular Surgery Interventional Anaemia Response (CAVIAR) Study: protocol for an observational cohort study to determine the impact and effect of preoperative anaemia management in cardiac and vascular surgical patients. BMJ Open. 2017 Apr 18;7(4):e014872. doi: 10.1136/bmjopen-2016-014872. PMID 28420664
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31902590/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28420664/